CLINICAL TRIAL: NCT00675116
Title: A Single-Blind, Randomised, Placebo Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GW823296 After Once-Daily Repeated Oral Doses in Healthy Male and Female Subjects
Brief Title: GW823296 Repeat Dose Study In Healthy Male And Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110371
Record Dates: First submitted 2008-04-24; First posted 2008-05-08 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: safety,; healthy volunteers,; GW823296,; pharmacokinetics

INTERVENTIONS:
Drug: GW823296

SUMMARY:
This is a study to evaluate the safety, tolerability and pharmacokinetics of GW823296 following 28 days, once-daily repeat oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a Physician Responsible, based on a medical evaluation including history, physical examination, laboratory tests, cardiac monitoring. A subject with a clinical abnormality or laboratory variables outside the reference range for the population being studied, with the exception of liver transaminases, troponin I and TSH, may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures. Please note that subjects should have liver transaminases, troponin I and TSH values within the range specified in the exclusion criteria below.
* Male or female between 18 and 65 years of age inclusive.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea and confirmed by screening follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml or <140 pmol/L.. Females on hormone replacement therapy (HRT) must discontinue HRT and their post-menopausal status confirmed as per above tests prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they are not allowed to use HRT during the study.
  * Child-bearing potential and agrees to use one of the contraception methods as per protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until at least 7 days after the last dose of study medication.
* Male subjects must agree to use one of the contraception methods as per protocol. This criterion must be followed from the time of the first dose of study medication until at least 7 days post last dose.
* No co-morbid Psychiatric Disorders as defined using the Mini International Neuropsychiatric Interview (M.I.N.I) scale.
* Normal neurological examination performed by the study neurologist
* A 12-lead ECG at screening showing no abnormalities that in the opinion of the Principal Investigator will compromise safety in this study.
* Body weight >/ 50 kg and BMI within the range 19.0 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject must be able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject
* The subject is available to complete the study

Exclusion Criteria:

* As a result of any of the medical interview, physical examination or screening investigations the Physician Responsible considers the subject unfit for the study.
* The subject or his/her family has a history of a drug or other allergy which in the opinion of the Physician Responsible contraindicates the participation in the study.
* Subjects with an unstable medical disorder or a disorder that would likely interfere with the action, absorption, distribution, metabolism or excretion of GW823296, may pose a safety concern, or interfere with accurate assessment of safety.
* The subject has a current or recent (within six months) documented gastrointestinal disease; a history of malabsorption, oesophageal reflux, or irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn, or any surgical intervention (e.g. cholecystectomy) which would be expected to influence the absorption of drugs.
* History of psychiatric illness
* Any history of a clinically significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer)
* The subject has screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5x upper limit of the normal range (ULN); testing may be repeated once to see if value returns to within acceptance range but any such laboratory abnormality must be resolved by the baseline visit.
* Subjects with a troponin I value >0.03 ng/mL at screening are not eligible. Testing may not be repeated. The subject should be referred to the treating physician for further evaluation, as appropriate.
* Subjects with a TSH value above the upper limit of the normal range (ULN) at screening are not eligible. The subject should be referred to the treating physician for further evaluation, as appropriate. Testing may be repeated once to see whether the value returns to within normal range but such abnormality must be resolved before the baseline visit.
* Subjects with a history of myopathy or rhabdomyolysis
* The subject is unable to abstain from strenuous physical activity for 72 hours prior to screening, for 72 hours prior first dosing until the last PK sample has been collected, and for 72 hours prior to the follow-up visit.
* The subject has donated a unit of blood (450 mL) within the previous 60 days or intends to donate in the month after completing the study
* Subjects with a history of eye disease (excluding moderate myopia) or clinically relevant eye examination finding, which in the opinion of the study ophthalmologist contraindicates their participation in the study
* The subjects is currently taking regular (or a course of) medication whether prescribed or not, including vitamins and herbal remedies, such as St John's Wort. Any concurrent medication will not be permitted for 48 hours before admission to the CPRU until the end of the study period (follow-up visit), unless in the opinion of the Investigator and the GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females).

[NOTE: 1 unit = 240mL beer, 90mL wine, or 30mL hard liquor]

* History of regular use of tobacco or nicotine containing products within 3 months prior to screening or a positive urine cotinine test result indicative of smoking at screening.
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV-1/2.
* The subject has a past history of drug/alcohol abuse or has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids, Benzodiazepines and Ethanol.
* Male subject intends to father a child during the study and the 3 months following the study
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing
* Lactating females
* Vulnerable subject (e.g. kept in detention)
* Subjects who have a history of hypersensitivity or intolerance to any of the study medications, or components thereof or other NK1 antagonists or history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor contraindicates their participation.
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events, Concomitant Medication,

SECONDARY OUTCOMES:
Physical Examination, Neurological Examination, Eye Examination, 12-lead ECG, Vital Signs, Laboratory Parameters, Pharmacokinetic Parameters

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia